CLINICAL TRIAL: NCT04546113
Title: Erector Spinae Plane Block Versus Paravertebral Block for Analgesic Outcomes After Cardiac Surgery (PEPS): a Prospective Randomized Comparative Study.
Brief Title: Erector Spinae Plane Block Versus Paravertebral Block for Analgesia After Cardiac Surgery (PEPS)
Acronym: PEPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Mutualiste Montsouris (Other)
Collaborators: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ANEST-03-2019
Record Dates: First submitted 2020-07-22; First posted 2020-09-11 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Pain Syndrome; Analgesia; Anesthesia, Local
Keywords: Cardiac surgery; Regional analgesia; Pain control
MeSH Terms: conditions — Somatoform Disorders; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paravertebral Block (Active Comparator): If the patient is randomized to group Paravertebral Block, the anesthesiologist performs TPVB after induction of general anesthesia. The patient is positioned in lateral decubitus position. The anesthetist performs the bilateral paravertebral block with ultrasound identification of the paravertebral space at the T4-T5 level. Slow injection of 0.3 to 0.35 ml / kg of ropivacaine on each side (diluted to 3.75 mg / ml = dilution in a 20 ml syringe with 10 ml of ropivacaine 7.5 mg / ml and 10 ml of NaCl 0.9%) after aspiration test.
  Interventions: Procedure: Ultrasound-guided Bilateral Paravertebral Block performed with a 20 ml injection of Ropivacaine 3,75 mg/ml/side
- Erector Spinae Plane Block (Experimental): If the patient is randomized to group "Erector Spinae Plane Block", the anesthesiologist performs the ESPb block after induction of general anesthesia. The patient is positioned in a right lateral decubitus position. The anesthesiologist performs the erector block of the spine ESP with ultrasound identification at the T4-T5 level (identify the 1st rib on ultrasound then the space T4 to T5). Slow injection of 20 ml of ropivacaine on each side (diluted to 3.75 mg / ml = dilution in a 20 ml syringe with 10 ml of ropivacaine 7.5 mg / ml and 10 ml of 0.9% NaCl) after aspiration test.
  The patient is then turned in left lateral decubitus position and the contralateral block is performed according to the same procedure.
  Interventions: Procedure: Ultrasound-guided Bilateral Erector Spinae plane Block performed with a 20 ml injection ropivacaine 3,75 mg/ml/side

INTERVENTIONS:
Procedure: Ultrasound-guided Bilateral Paravertebral Block performed with a 20 ml injection of Ropivacaine 3,75 mg/ml/side — Bilateral injection of 20 ml of Ropivacaine 3,75 mg/ml/side
  Arms: Paravertebral Block
Procedure: Ultrasound-guided Bilateral Erector Spinae plane Block performed with a 20 ml injection ropivacaine 3,75 mg/ml/side — Bilateral injection of 20 ml of Ropivacaine 3,75 mg/ml/side
  Arms: Erector Spinae Plane Block

SUMMARY:
The purpose of this randomized double-blind study is to compare the analgesic efficacy of the bilateral Erector Spinae Plane (ESP) block versus the bilateral Thoracic Paravertebral block (TPVB), by ultrasound-guided single injection in patients who underwent sternotomy for cardiac surgery.

DETAILED DESCRIPTION:
Cardiac surgery causes moderate to severe postoperative pain during the first 24 - 48 post-operative hours. This pain is greatly increased by mobilization (respiratory physiotherapy) and leads to the consumption of morphine.

Appropriate analgesia, along with a reduction in morphine consumption are important factors in reducing morbidity after cardiac surgery and allow better postoperative rehabilitation.

Recently, the concept of multimodal analgesia has become established, which corresponds to ensuring optimal analgesia through the use of non-morphine drugs associated with locoregional analgesia.

During cardiac surgery, Paravertebral block (TPVB) technique is the first line of reference in our establishment. Lately, a new approach of blocking the intercostal nerves called Erector Spinae Plane block (ESP) has been discovered. It is a technique that seems simpler and safer than TPVB.

Until now, the analgesic efficacy of the ESP block compared to TPVB after cardiac surgery by sternotomy has never been studied.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing any (scheduled) surgery of the heart (valve or coronary surgery) via a median sternotomy
* Physical status classification (ASA) ≤3
* Patients benefiting from a Social Security scheme or benefiting from it through a third party

Exclusion Criteria:

* Emergency cardiac surgery
* Exclusion criteria related to cardiac surgery with thoracotomy, occurrence of aortic dissection, redo surgery.
* Aortic counterpulsation
* Preoperative cardiogenic shock
* LVEF< 30%
* Severe preoperative chronic or acute renal failure with creatinine clearance less than 30 mL / min according to the MDRD formula
* Pre-existing psychiatric pathology, including addiction to opioids
* Physical or intellectual incapacity to use a PCA
* Known allergy or hypersensitivity to any of the study drugs or analgesia protocol (ropivacaine, paracetamol, opioids)
* Contraindication for performing the paravertebral block and Erector of the spine (ESP): Infection at the site of injection, severe hemostasis disorder, thoracic spinal pathology making the procedure difficult or dangerous to operate
* Obese patient (BMI> 30kg / m2) with poorly perceived thoracic spinous processes.
* vulnerable patients(Pregnant or breastfeeding women, persons benefiting from enhanced protection, namely persons deprived of their liberty by a judicial or administrative decision, adults under legal protection).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Pain assessment | 6 hours from the end of the surgery
  Pain assessment measured with Visual Analogue Scale (VAS) between 0 (no pain, best outcome) and 10 (worst possible pain, worst outcome) at mobility, (respiratory effort during peak flow meter measurement)

SECONDARY OUTCOMES:
Efficacy of the block (a) | During the surgery
  Based on hemodynamic response to incision and sternotomy (increase in heart rate, measured in beats per minute (bpm)
Efficacy of the block (b) | During the surgery
  Based on variations in the ANI (Anti Nociceptive Index) value (scale from 0 (maximum of nociception) to 100 (complete analgesia))
Efficacy of the block (c) | During the surgery
  Based on hemodynamic response to incision and sternotomy (increase in blood pressure, measured in mmHg). Blood pressure numbers of less than 120/80 mm Hg are considered within the normal range.
Intraoperative sufentanil consumption | During the surgery
  Intraoperative sufentanil consumption (at the discretion of physicians based on haemodynamic variations and ANI values). Measured in ng/ml.
Postoperative pain assessment | 3, 6, 12, 24, 48 hours from the end of the surgery
  Pain assessment measured with Visual Analogue Scale between 0 (no pain, best outcome) and 10 (worst possible pain and and worst outcome) at mobility, (respiratory effort during peak flow meter measurement)
Postoperative Morphine consumption | 3, 6, 12, 24, 48 hours from the end of the surgery
  Morphine PCA consumption, measured in mg/h.
Side effects associated to morphine | 3, 6, 12, 24, 48 hours from the end of the surgery
  Incidence of post operative nausea, vomiting and sedation
Complication(s) associated to the procedure | 48 hours from the end of the surgery
  Pneumothorax, major hematoma, sympathetic block

CONTACTS AND LOCATIONS:
Overall Officials: Olivier MONTANDRAU, MD, Principal Investigator — Institut Mutualiste Montsouris
Locations (1):
- Institut Mutualiste montsouris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Montandrau O, Kattou F, Arana H, Rekik M, Ait Hamou N, Weisslinger SJ, Teil E, Mekaouar S, Bargaoui A, Bouattour K, Bey Boumezrag C, Lacombe JM, Lebatard N, Zannis K, Beaussier M. Ultrasound-guided thoracic paravertebral block versus erector spinae plane block analgesia for cardiac surgery with median sternotomy: a noninferiority randomised controlled trial. Br J Anaesth. 2026 Feb;136(2):687-694. doi: 10.1016/j.bja.2025.10.039. Epub 2025 Nov 24. PMID 41290467